CLINICAL TRIAL: NCT00935727
Title: Pilot Study to Define Parameters of Elastography Compared to Color Flow Doppler Ultrasound in Renal Transplants
Brief Title: Elastographic Imaging of Renal Transplants
Acronym: Elastorenal
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: images obtained were non-diagnostic
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Memorial Hermann Hospital (Other)
Responsible Party: Alan Cohen, MD, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-06-0255
Record Dates: First submitted 2009-05-08; First posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Renal Transplant
Keywords: renal transplant; ultrasound; elastography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): normally functioning transplanted kidneys
  Interventions: Other: Elastographic imaging
- 2 (Other): transplanted kidney undergoing known rejection or other known abnormality
  Interventions: Other: Elastographic imaging
- 3 (Other): transplanted kidney with unknown diagnosis
  Interventions: Other: Elastographic imaging

INTERVENTIONS:
Other: Elastographic imaging — ultrasound imaging using a specialized computer that processes the data for tissue hardness

SUMMARY:
The study was developed to acquire images of normal, then abnormal, then unknown diagnosis for transplanted kidneys in order to determine whether the elastography imaging modality, a type of ultrasound imaging, can provide data useful for diagnosis of renal transplant abnormalities.

The specific aims of this study are:

1. To define normal elastography imaging by correlation with clinical findings.
2. To define specific abnormal elastography images by correlation with clinical findings.
3. To determine whether elastography could be useful in early diagnosis of abnormalities of renal transplants, especially in early rejection.

DETAILED DESCRIPTION:
The study is collecting standard ultrasound and elastographic images of transplanted kidneys in order to perfect the imaging technique to get the best pictures, and to evaluate these images for characteristics that may be of diagnostic value.

ELIGIBILITY:
Inclusion Criteria:

* Adult (over 18) male or female renal transplant patient
* normally functioning
* or being evaluated for a possible problem

Exclusion Criteria:

* unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Identification of features of a set of elastography images that can be characterized as those of a normally functioning transplanted kidney, or those of specific abnormalities | after up to 50 "normal" images are collected

SECONDARY OUTCOMES:
Assessment of the value of renal transplant imaging by elastography compared to standard ultrasound | by the time up to 100 images are obtained

CONTACTS AND LOCATIONS:
Overall Officials: Alan M Cohen, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Jonathan Ophir, PhD, Study Director — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Background] Weitzel WF, Kim K, Rubin JM, Xie H, O'Donnell M. Renal advances in ultrasound elasticity imaging: measuring the compliance of arteries and kidneys in end-stage renal disease. Blood Purif. 2005;23(1):10-7. doi: 10.1159/000082005. PMID 15627731
- See also: general information about elastography — http://www.elastography.com